CLINICAL TRIAL: NCT05676255
Title: The SUPORT Project: Leveraging Social Connection by Including Informal Caregivers in an Internet Video Conference-based Compassion Meditation Intervention to Reduce Psychological Distress in Breast Cancer Survivors
Brief Title: The Breast Cancer Survivors and Partners Online Research Together (SUPORT) Project
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Thaddeus Pace, Associate Professor of Nursing, Psychiatry, and Psychology, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: STUDY00001225; R01CA264047 (NIH)
Record Dates: First submitted 2022-12-22; First posted 2023-01-09 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer Female; Psychological Distress

STUDY DESIGN:
Intervention Model Description: randomized clinical trial design
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants will be informed of their group assignment only after completion of the baseline (T1) assessment, and data collectors will be blinded to study group assignment for all future assessments. Participants will be asked to not discuss their group assignment with anyone other than the study coordinator. The PI and other investigators will be blinded to arm assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cognitively-Based Compassion Training for Survivors (CBCT-S) (Experimental): CBCT-S is a secular adaptation of techniques derived from traditional Tibetan Buddhist methods for cultivating compassion known as lo-jong. CBCT-S will be administered to breast cancer survivors and will not including supportive partners.
  Module 1 (Week 1): Overview and Connecting to A Moment of Nurturance
  Module 2 (Week 2) Developing Stable and Clear Attention
  Module 3 (Week 3): Enhancing Self Awareness
  Module 4 (Week 4): Cultivating Self compassion Part 1: Accepting our Suffering
  Module 5 (Week 5): Self Compassion Part 2: Finding Meaning in Suffering.
  Module 6(Week 6): Expanding our Circle of Concern
  Module 7 (Week 7): Deepening Gratitude and Tenderness
  Module 8 (Week 8): Harnessing the Power of Compassion
  Interventions: Behavioral: Cognitively-Based Compassion Training for Survivors
- Cognitively-Based Compassion Training for Dyads (CBCT-D) (Experimental): CBCT-D is a secular adaptation of techniques derived from traditional Tibetan Buddhist methods for cultivating compassion known as lo-jong. CBCT-D will be administered to breast cancer survivors and supportive partners together.
  Module 1 (Week 1): Overview and Connecting to A Moment of Nurturance
  Module 2 (Week 2) Developing Stable and Clear Attention
  Module 3 (Week 3): Enhancing Self Awareness
  Module 4 (Week 4): Cultivating Self compassion Part 1: Accepting our Suffering
  Module 5 (Week 5): Self Compassion Part 2: Finding Meaning in Suffering.
  Module 6(Week 6): Expanding our Circle of Concern
  Module 7 (Week 7): Deepening Gratitude and Tenderness
  Module 8 (Week 8): Harnessing the Power of Compassion
  Interventions: Behavioral: Cognitively-Based Compassion Training for Dyads
- Health Education (Active Comparator): HE focuses on topics relevant to health and cancer, but is also intended for individuals who are not cancer survivors themselves.
  HE will be administered to both breast cancer survivors and supportive partners together.
  Module I (Week 1): Cancer Advocacy.
  Module II (Week 2): Health Through the Lifespan.
  Module III (Week 3): Nutrition.
  Module III (Week 4): Nutrition.
  Module IV (Week 5): Physical Activity.
  Module V (Week 6): Sleep.
  Module VI (Week 7): Stress.
  Module VII (Week 8): Mental Health and Social Support.
  Interventions: Behavioral: Health Education

INTERVENTIONS:
Behavioral: Cognitively-Based Compassion Training for Survivors — CBCT-S is a secular adaptation of techniques derived from traditional Tibetan Buddhist methods for cultivating compassion known as lo-jong. CBCT-S will be administered to breast cancer survivors and will not including supportive partners.
  Module 1 (Week 1): Overview and Connecting to A Moment of Nurturance
  Module 2 (Week 2) Developing Stable and Clear Attention
  Module 3 (Week 3): Enhancing Self Awareness
  Module 4 (Week 4): Cultivating Self compassion Part 1: Accepting our Suffering
  Module 5 (Week 5): Self Compassion Part 2: Finding Meaning in Suffering.
  Module 6(Week 6): Expanding our Circle of Concern
  Module 7 (Week 7): Deepening Gratitude and Tenderness
  Module 8 (Week 8): Harnessing the Power of Compassion
  Other Names: CBCT-S
  Arms: Cognitively-Based Compassion Training for Survivors (CBCT-S)
Behavioral: Cognitively-Based Compassion Training for Dyads — CBCT-D is a secular adaptation of techniques derived from traditional Tibetan Buddhist methods for cultivating compassion known as lo-jong. CBCT-D will be administered to breast cancer survivors and supportive partners together.
  Module 1 (Week 1): Overview and Connecting to A Moment of Nurturance
  Module 2 (Week 2) Developing Stable and Clear Attention
  Module 3 (Week 3): Enhancing Self Awareness
  Module 4 (Week 4): Cultivating Self compassion Part 1: Accepting our Suffering
  Module 5 (Week 5): Self Compassion Part 2: Finding Meaning in Suffering.
  Module 6(Week 6): Expanding our Circle of Concern
  Module 7 (Week 7): Deepening Gratitude and Tenderness
  Module 8 (Week 8): Harnessing the Power of Compassion
  Other Names: CBCT-D
  Arms: Cognitively-Based Compassion Training for Dyads (CBCT-D)
Behavioral: Health Education — HE focuses on topics relevant to health and cancer, but is also intended for individuals who are not cancer survivors themselves.
  HE will be administered to both breast cancer survivors and supportive partners together.
  Module I (Week 1): Cancer Advocacy.
  Module II (Week 2): Health Through the Lifespan.
  Module III (Week 3): Nutrition.
  Module III (Week 4): Nutrition.
  Module IV (Week 5): Physical Activity.
  Module V (Week 6): Sleep.
  Module VI (Week 7): Stress.
  Module VII (Week 8): Mental Health and Social Support.
  Other Names: HE
  Arms: Health Education

SUMMARY:
Many breast cancer survivors (estimated 70% in some studies) experience clinically significant depression and/or anxiety in the months and years after finishing cancer treatments. This research will build on the rigor of prior research to reduce breast cancer survivor depression and anxiety with a compassion meditation intervention called CBCT (Cognitively-Based Compassion Training) for online synchronous delivery that is also inclusive of informal caregivers (i.e., adult family members who live with and typically provide half the care for survivors, aka supportive partners).

DETAILED DESCRIPTION:
The goal of this project is to determine if CBCT (Cognitively-Based Compassion Training) can reduce distress for survivors compared to an attention control (Health Education; HE) when delivered by Zoom to both survivors and caregivers/ supportive partners as a dyad (i.e., CBCT for dyads; CBCT-D). We will also test whether instructing survivors and caregivers/ supportive partners together in CBCT (CBCT-D) reduces distress more than when survivors receive CBCT instruction by themselves, without caregivers/ supportive partners (i.e., CBCT for survivors; CBCT-S). The following specific aims address these questions:

Aim 1: Determine if survivors and caregivers/ supportive partners exhibit less depression and anxiety (primary outcomes) when survivors receive online CBCT along with their informal caregiver// supportive partner (CBCT-D), compared to when survivors receive online CBCT alone (CBCT-S) or when survivors and informal caregivers// supportive partners receive online HE. We will recruit dyads (N=226) consisting of survivors (between 3 months and 5 years post treatments with curative intent, i.e., chemotherapy, radiation, surgery) and their caregivers/ supportive partners. H1: Survivors and caregivers randomized to CBCT-D will exhibit greater improvements in distress (i.e., depression, anxiety; primary outcomes in survivors) at months 2, 3, and 8 versus those randomized to CBCT-S or HE.

Aim 2: Test the extent to which reductions in survivor's depression and anxiety from online CBCT-D are mediated by social connection, dyadic function, and caregiver/ supportive partner distress. H2a: Survivor's social connection and dyadic function will mediate the effects of online CBCT-D versus HE on survivor's distress at months 2, 3 and 8. H2b: Caregiver's social connection, dyadic function, and distress will mediate the effects of CBCT-D versus CBCT-S or HE on survivor's distress.

Aim 3: Explore the effects of online CBCT-D versus CBCT-S and HE on survivor diurnal cortisol rhythm at months 2, 3 and 8, and the extent to which cortisol rhythm is a marker versus mediator of improvements in survivor's distress at month 2, 3, and 8.

ELIGIBILITY:
Breast cancer survivors:

Inclusion Criteria:

* biological sex: woman
* able to speak and understand English
* have a diagnosis of a breast cancer
* have completed primary curative cancer treatments (i.e., surgery, radiation, chemotherapy) except for hormonal therapies (e.g., aromatase inhibitors) or trastuzumab a minimum of 3 months and a maximum of 5 years before starting CBCT or the control
* have a supportive partner (aka caregiver) who can participate with them

Exclusion Criteria:

* nursing home resident
* have ongoing (1 or more meditation sessions per week) or past regular meditation experience in the last 4 years (i.e., more than two meditation sessions [completed or attempted] per year, either with a group or individually, to be evaluated by the Principal Investigator)

Supportive partners (aka informal caregivers)

Inclusion Criteria:

* named by the survivor
* live in the same household as the survivor
* able to speak and understand English

Exclusion Criteria:

* have ongoing (1 or more meditation sessions per week) or past regular meditation experience in the last 4 years (i.e., more than two meditation sessions [completed or attempted] per year, either with a group or individually, to be evaluated by the Principal Investigator)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 452 (Estimated)
Dates: Start 2023-03-20 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Change in depression features | Change from baseline depression to 8 weeks after the start of intervention
  The difference in the change in depression features between the intervention arms from before to 8 weeks after start of the interventions will be measured with the Patient-Reported Outcomes Measurement Information System short form Depression - 8a.
Change in anxiety features | Change from baseline anxiety to 8 weeks after the start of intervention
  The difference in the change in anxiety features between the intervention arms from before to 8 weeks after start of the interventions will be measured with the Patient-Reported Outcomes Measurement Information System short form Anxiety - 8a.

SECONDARY OUTCOMES:
Change in depression features | Change from baseline depression to 12 weeks after the start of intervention
  The difference in the change in depression features between the intervention arms from before to 12 weeks after start of the interventions will be measured with the Patient-Reported Outcomes Measurement Information System short form Depression - 8a.
Change in anxiety features | Change from baseline anxiety to 12 weeks after the start of intervention
  The difference in the change in anxiety features between the intervention arms from before to 12 weeks after start of the interventions will be measured with the Patient-Reported Outcomes Measurement Information System short form Anxiety - 8a.
Change in depression features | Change from baseline depression to 32 weeks after the start of intervention
  The difference in the change in depression features between the intervention arms from before to 32 weeks after start of the interventions will be measured with the Patient-Reported Outcomes Measurement Information System short form Depression - 8a.
Change in anxiety features | Change from baseline anxiety to 32 weeks after the start of intervention
  The difference in the change in anxiety features between the intervention arms from before to 32 weeks after start of the interventions will be measured with the Patient-Reported Outcomes Measurement Information System short form Anxiety - 8a.

CONTACTS AND LOCATIONS:
Overall Officials: Thaddeus Pace, PhD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
not applicable as of current version date